CLINICAL TRIAL: NCT04603118
Title: Comparison of Optic Nerve Sheath Diameters Measured by Optic Ultrasonography Before and After Lumbar Puncture in Idiopathic Intracranial Hypertension Patients
Brief Title: Optic Nerve Sheath Diameters in Idiopathic Intracranial Hypertension Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Zehra Bozdoğan Şenel, Medical Doctor, Principal Investigator, Ege University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DIA-SONSD
Record Dates: First submitted 2020-10-03; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Pseudotumor Cerebri
Keywords: Idiopathic intracranial hypertension; Optic nerve sheath diameter measurement; Increased intracranial pressure; Lumbar puncture
MeSH Terms: conditions — Pseudotumor Cerebri; Intracranial Hypertension | interventions — Spinal Puncture

STUDY DESIGN:
Intervention Model Description: Patients who applied to the neurology clinics and were diagnosed with IIH were included in the study. The control group consisted of 22 individuals who applied with other complaints than headaches. ONSD was measured from both eyes before and after the LP. After pre-LP measurements were taken, opening and closing cerebrospinal fluid pressure was measured. In the control group, ONSD was measured with optic USG.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The patients with Idiopathic intracranial hypertension (IIH) (Other): 33 patients who applied to the neurology clinic with the pre-diagnosis of IIH were performed lumbar puncture. 25 of them diagnosed with IIH. Optic nerve sheath diameter was measured by optic ultrasonography from both eyes before and after the LP.
  Interventions: Procedure: Optic ultrasonography; Procedure: Lumbar puncture
- Control group (Other): In the control group, optic nerve sheath diameter was measured from both eyes by optic ultrasonography.
  Interventions: Procedure: Optic ultrasonography

INTERVENTIONS:
Procedure: Optic ultrasonography
Procedure: Lumbar puncture
  Arms: The patients with Idiopathic intracranial hypertension (IIH)

SUMMARY:
Idiopathic intracranial hypertensionis a type of increased intracranial pressure. Diagnosis is made by lumbar puncture, which is an invasive technique. The relationship between ICP and optic nerve sheath diameters (ONSD) were examined in our study. Thus, it was investigated whether the optic nerve sheath diameter could be used in the diagnosis of IIH. In the present study, it was found that ONSD measurement by optic USG significantly reflects increased ICP and decreasing pressure via LP is rapidly reflects to ONSD measurement. And it is suggested that ONSD measurements by optic USG, a non-invasive method, can be used in the diagnosis and follow-up of IIH patients.

DETAILED DESCRIPTION:
Backgrounds: Idiopathic intracranial hypertension (IIH); symptoms include headaches, blurred vision and papilledema which may lead to permanent visual loss. Definitive diagnosis of IIH usually requires the measurement of intracranial pressure (ICP) via lumbar puncture (LP) which is an invasive technique. In our study, the relationship between ICP and optic nerve sheath diameters (ONSD) were examined. Thus it was investigated whether optic nerve ultrasonography (USG) is a useful tool instead of LP for the diagnosis of IIH.

Methods: A total of 25 patients who applied to the neurology clinics of Ankara Numune Training and Research Hospital between May 2014 and December 2015 and were diagnosed with IIH were included in the study. The control group consisted of 22 individuals who applied with other complaints than headaches. ONSD was measured from both eyes before and after the LP. After pre-LP measurements were taken, opening and closing CSF (cerebrospinal fluid) pressure was measured. In the control group, ONSD was measured with optic USG.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic intracranial hypertension
* Adults aged 17-65

Exclusion Criteria:

* In cranial imaging, if pathology such as tumor, sinus vein thrombosis is detected
* People for whom lumbar puncture is contraindicated or cannot be performed

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-04-01 (Actual)

PRIMARY OUTCOMES:
Correlation between intracranial pressure change and optic nerve sheath diameter | Baseline to 10-15 minutes after lumbar puncture
  Before and after lumbar puncture, optic nerve sheath diameter measured with optic ultrasonography. The correlation of these measurements with cerebrospinal fluid opening and closing pressures was investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Oğuzhan Kurşun, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Numune Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
For a reasonable purpose, data can be given to appropriate people if desired.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data is available for one year after publication
Access Criteria: The reason and purpose of the request is clearly explained and the appropriate persons can access it via e-mail.

REFERENCES:
- [Background] Soler D, Cox T, Bullock P, Calver DM, Robinson RO. Diagnosis and management of benign intracranial hypertension. Arch Dis Child. 1998 Jan;78(1):89-94. doi: 10.1136/adc.78.1.89. No abstract available. PMID 9534686
- [Background] Sorensen PS, Krogsaa B, Gjerris F. Clinical course and prognosis of pseudotumor cerebri. A prospective study of 24 patients. Acta Neurol Scand. 1988 Feb;77(2):164-72. doi: 10.1111/j.1600-0404.1988.tb05888.x. PMID 3364156
- [Background] Wall M, George D. Idiopathic intracranial hypertension. A prospective study of 50 patients. Brain. 1991 Feb;114 ( Pt 1A):155-80. PMID 1998880
- [Background] Giuseffi V, Wall M, Siegel PZ, Rojas PB. Symptoms and disease associations in idiopathic intracranial hypertension (pseudotumor cerebri): a case-control study. Neurology. 1991 Feb;41(2 ( Pt 1)):239-44. doi: 10.1212/wnl.41.2_part_1.239. PMID 1992368
- [Background] Durcan FJ, Corbett JJ, Wall M. The incidence of pseudotumor cerebri. Population studies in Iowa and Louisiana. Arch Neurol. 1988 Aug;45(8):875-7. doi: 10.1001/archneur.1988.00520320065016. PMID 3395261
- [Background] Dhungana S, Sharrack B, Woodroofe N. Idiopathic intracranial hypertension. Acta Neurol Scand. 2010 Feb;121(2):71-82. doi: 10.1111/j.1600-0404.2009.01172.x. Epub 2009 Nov 23. PMID 19930211
- [Background] Radhakrishnan K, Ahlskog JE, Garrity JA, Kurland LT. Idiopathic intracranial hypertension. Mayo Clin Proc. 1994 Feb;69(2):169-80. doi: 10.1016/s0025-6196(12)61045-3. PMID 8309269
- [Background] Degnan AJ, Levy LM. Pseudotumor cerebri: brief review of clinical syndrome and imaging findings. AJNR Am J Neuroradiol. 2011 Dec;32(11):1986-93. doi: 10.3174/ajnr.A2404. Epub 2011 Jun 16. PMID 21680652
- [Background] Brazis PW. Clinical review: the surgical treatment of idiopathic pseudotumour cerebri (idiopathic intracranial hypertension). Cephalalgia. 2008 Dec;28(12):1361-73. doi: 10.1111/j.1468-2982.2008.01778.x. PMID 19037972
- [Background] Levine DN. Ventricular size in pseudotumor cerebri and the theory of impaired CSF absorption. J Neurol Sci. 2000 Aug 15;177(2):85-94. doi: 10.1016/s0022-510x(00)00348-8. PMID 10980304
- [Background] Bruce BB, Kedar S, Van Stavern GP, Monaghan D, Acierno MD, Braswell RA, Preechawat P, Corbett JJ, Newman NJ, Biousse V. Idiopathic intracranial hypertension in men. Neurology. 2009 Jan 27;72(4):304-9. doi: 10.1212/01.wnl.0000333254.84120.f5. Epub 2008 Oct 15. PMID 18923135
- [Background] Avery RA, Shah SS, Licht DJ, Seiden JA, Huh JW, Boswinkel J, Ruppe MD, Chew A, Mistry RD, Liu GT. Reference range for cerebrospinal fluid opening pressure in children. N Engl J Med. 2010 Aug 26;363(9):891-3. doi: 10.1056/NEJMc1004957. No abstract available. PMID 20818852
- [Background] Hayreh SS. Pathogenesis of optic disc edema in raised intracranial pressure. Prog Retin Eye Res. 2016 Jan;50:108-44. doi: 10.1016/j.preteyeres.2015.10.001. PMID 26453995
- [Background] Hayreh SS. Optic disc edema in raised intracranial pressure. V. Pathogenesis. Arch Ophthalmol. 1977 Sep;95(9):1553-65. doi: 10.1001/archopht.1977.04450090075006. PMID 71138
- [Background] Suzuki H, Takanashi J, Kobayashi K, Nagasawa K, Tashima K, Kohno Y. MR imaging of idiopathic intracranial hypertension. AJNR Am J Neuroradiol. 2001 Jan;22(1):196-9. PMID 11158909
- [Background] Brodsky MC, Vaphiades M. Magnetic resonance imaging in pseudotumor cerebri. Ophthalmology. 1998 Sep;105(9):1686-93. doi: 10.1016/S0161-6420(98)99039-X. PMID 9754178
- [Result] Girisgin AS, Kalkan E, Kocak S, Cander B, Gul M, Semiz M. The role of optic nerve ultrasonography in the diagnosis of elevated intracranial pressure. Emerg Med J. 2007 Apr;24(4):251-4. doi: 10.1136/emj.2006.040931. PMID 17384377
- [Result] Le A, Hoehn ME, Smith ME, Spentzas T, Schlappy D, Pershad J. Bedside sonographic measurement of optic nerve sheath diameter as a predictor of increased intracranial pressure in children. Ann Emerg Med. 2009 Jun;53(6):785-91. doi: 10.1016/j.annemergmed.2008.11.025. Epub 2009 Jan 23. PMID 19167786
- [Result] Geeraerts T, Duranteau J, Benhamou D. Ocular sonography in patients with raised intracranial pressure: the papilloedema revisited. Crit Care. 2008;12(3):150. doi: 10.1186/cc6893. Epub 2008 May 16. PMID 18495051
- [Result] Soldatos T, Karakitsos D, Chatzimichail K, Papathanasiou M, Gouliamos A, Karabinis A. Optic nerve sonography in the diagnostic evaluation of adult brain injury. Crit Care. 2008;12(3):R67. doi: 10.1186/cc6897. Epub 2008 May 13. PMID 18477382
- [Result] Tayal VS, Neulander M, Norton HJ, Foster T, Saunders T, Blaivas M. Emergency department sonographic measurement of optic nerve sheath diameter to detect findings of increased intracranial pressure in adult head injury patients. Ann Emerg Med. 2007 Apr;49(4):508-14. doi: 10.1016/j.annemergmed.2006.06.040. Epub 2006 Sep 25. PMID 16997419
- [Result] Blaivas M, Theodoro D, Sierzenski PR. Elevated intracranial pressure detected by bedside emergency ultrasonography of the optic nerve sheath. Acad Emerg Med. 2003 Apr;10(4):376-81. doi: 10.1111/j.1553-2712.2003.tb01352.x. PMID 12670853
- [Result] Rajajee V, Vanaman M, Fletcher JJ, Jacobs TL. Optic nerve ultrasound for the detection of raised intracranial pressure. Neurocrit Care. 2011 Dec;15(3):506-15. doi: 10.1007/s12028-011-9606-8. PMID 21769456
- [Result] Kimberly HH, Shah S, Marill K, Noble V. Correlation of optic nerve sheath diameter with direct measurement of intracranial pressure. Acad Emerg Med. 2008 Feb;15(2):201-4. doi: 10.1111/j.1553-2712.2007.00031.x. PMID 18275454
- [Result] Dubost C, Le Gouez A, Jouffroy V, Roger-Christoph S, Benhamou D, Mercier FJ, Geeraerts T. Optic nerve sheath diameter used as ultrasonographic assessment of the incidence of raised intracranial pressure in preeclampsia: a pilot study. Anesthesiology. 2012 May;116(5):1066-71. doi: 10.1097/ALN.0b013e318246ea1a. PMID 22258019
- [Result] Amini A, Kariman H, Arhami Dolatabadi A, Hatamabadi HR, Derakhshanfar H, Mansouri B, Safari S, Eqtesadi R. Use of the sonographic diameter of optic nerve sheath to estimate intracranial pressure. Am J Emerg Med. 2013 Jan;31(1):236-9. doi: 10.1016/j.ajem.2012.06.025. Epub 2012 Aug 31. PMID 22944553
- [Result] Bauerle J, Nedelmann M. Sonographic assessment of the optic nerve sheath in idiopathic intracranial hypertension. J Neurol. 2011 Nov;258(11):2014-9. doi: 10.1007/s00415-011-6059-0. Epub 2011 Apr 28. PMID 21523461
- [Result] Dubourg J, Javouhey E, Geeraerts T, Messerer M, Kassai B. Ultrasonography of optic nerve sheath diameter for detection of raised intracranial pressure: a systematic review and meta-analysis. Intensive Care Med. 2011 Jul;37(7):1059-68. doi: 10.1007/s00134-011-2224-2. Epub 2011 Apr 20. PMID 21505900
- [Result] Roque PJ, Wu TS, Barth L, Drachman D, Khor KN, Lovecchio F, Stapczynski S. Optic nerve ultrasound for the detection of elevated intracranial pressure in the hypertensive patient. Am J Emerg Med. 2012 Oct;30(8):1357-63. doi: 10.1016/j.ajem.2011.09.025. Epub 2011 Dec 26. PMID 22204998

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT04603118/Prot_SAP_000.pdf